CLINICAL TRIAL: NCT02856269
Title: Zinc Supplementation and Cardiovascular Risk in HIV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Grace McComsey (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor-Investigator, Grace McComsey, MD, University Hospitals Cleveland Medical Center
Organization: University Hospitals Cleveland Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 02-15-07; 1R21AT009153-01 (NIH)
Record Dates: First submitted 2016-07-29; First posted 2016-08-04 (Estimated); Results first posted 2022-02-11 (Actual); Last update posted 2022-02-11 (Actual); Status verified 2022-02

CONDITIONS: HIV; Inflammation
Keywords: Zinc
MeSH Terms: conditions — Inflammation | interventions — gluconic acid

STUDY DESIGN:
Intervention Model Description: This is a pilot open labeled randomized double arm trial, studying zinc supplementation to prevent HIV comorbidities that are linked to inflammation. Patients will be given zinc gluconate 45 mg capsule once daily in one arm, and 90 mg zinc gluconate in the other arm for 16 weeks.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Patients and the research nurse are unblinded. The research assistant and the principle investigator are blinded.
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 45 mg daily (Active Comparator): Participants in this arm will take a daily 45 mg dose of zinc gluconate.
  Interventions: Dietary Supplement: Zinc gluconate
- 90 mg daily (Active Comparator): Participants in this arm will take a daily 90 mg dose of zinc gluconate.
  Interventions: Dietary Supplement: Zinc gluconate

INTERVENTIONS:
Dietary Supplement: Zinc gluconate — Participants will take a daily dose of zinc gluconate.

SUMMARY:
The purpose of this pilot study is to determine whether zinc supplementation significantly affects immune activation in HIV-infected subjects.

DETAILED DESCRIPTION:
Zinc is a dietary supplement with compelling preclinical evidence for potential health benefit that could be expanded not only to the entire HIV population, but also to other inflammatory conditions that share many facets of HIV infection, namely the persistent intestinal barrier dysfunction, monocyte activation and heightened inflammation state.

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 infection
* Age ≥18 years
* Zinc level ≤0.75 mg/L
* Receiving a stable antiretroviral regimen with no plans to change during study
* Documentation of an HIV-1 RNA level of ≤400 copies/mL
* No diarrhea or nausea/vomiting for the last month

Exclusion Criteria:

* Pregnancy/lactation
* Presence of inflammatory condition
* Regular use of agents that may affect inflammation in the last 3 months. The regular use of NSAIDS, aspirin, or statins will be allowed as long as dose has been stable for the last 3 months and is not expected to change during the study.
* Presence of active neoplastic diseases requiring chemotherapy and/or use of immunosuppressive drugs
* Known cardiovascular disease
* Uncontrolled diabetes
* Allergy or intolerance to zinc sulfate.
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) > 2.5 x Upper limit of normal (ULN)
* Hemoglobin < 9.0 g/dL
* glomerular filtration rate (GFR) < 50 mL/min

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2016-09; Primary Completion 2018-04-16 (Actual); Study Completion 2018-04-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Grace McComsey, MD, Principal Investigator — University Hospitals Cleveland Medical Center
Locations (1):
- University Hospitals Cleveland Medical Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited based on physician referral at University Hospitals Cleveland Medical Center between September 2016 and February 2018.
Pre-assignment Details: Of 118 patients screened, 52 met inclusion criteria and were randomized to treatment.
Period: Overall Study
Arm/Group | 45 mg Daily | 90 mg Daily
Started | 25 | 27
Completed | 24 | 24
Not Completed | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 45 mg Daily | 90 mg Daily | Total
Number analyzed (Participants) | 25 | 27 | 52
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 23 | 1 | 24
  >=65 years | 2 | 26 | 28
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 54 [48 to 60] | 47 [38 to 54.50] | 49 [38 to 60]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 7 | 12
  Male | 20 | 20 | 40
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 3 | 3
  Not Hispanic or Latino | 25 | 24 | 49
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 18 | 20 | 38
  White | 7 | 7 | 14
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 25 | 27 | 52
Zinc levels [Median (Inter-Quartile Range); unit: μg/dL] — Median and Inter-Quartile range of zinc blood levels in μg/dL
  μg/dL | 74.00 [64.00 to 83.00] | 73.00 [66.00 to 86.00] | 73 [64 to 86]

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Decreased Inflammation Markers sCD14, sTNF-RI, and High Sensitivity C Reactive Protein (Hs-CRP)
Description: Percentage of participants with the following inflammatory markers decrease (sCD14) Soluble cluster of differentiation 14, (sTNF-RI) soluble Tumor Necrosis Factor alpha receptor I, (hs-CRP) High sensitivity C-reactive protein. These inflammatory markers are measured in the blood by enzyme-linked immunoassay ELISA.
Time Frame: Baseline and 16 Weeks
Population: Intent to treat population (all participants assigned to zinc 45 mmg or zinc 90 mg).
Measure: Count of Participants; unit: Participants
Arm/Group | 45 mg Daily | 90 mg Daily
Number analyzed (Participants) | 25 | 27
Participants
  sCD14 | 15 | 15
  sTNF-RI | 14 | 15
  hs-CRP | 12 | 15
Statistical Analysis 1: Comparison: 45 mg Daily vs 90 mg Daily; Test type: Other — Wilcoxon rank sum tests, X2 tests, Fisher exact tests, Kolmogorov-Smirnov; Cohen's D value = 0.8 — The Cohen's d is calculated after Box-Cox transformation. Small effect <= 0.2, Medium effect [0.3, 0.8]; Large effect >0.8

2. Secondary Outcome: Percentage of Participants That Reached the Zinc Sufficient Level After Treatment
Description: After treatment, zinc was measured in the blood. Patients are considered sufficient if zinc levels >75 μg/dL.
Time Frame: 16 Weeks
Measure: Number; unit: percentage of participants
Arm/Group | 45 mg Daily | 90 mg Daily
Number analyzed (Participants) | 25 | 27
percentage of participants | 88 | 96

ADVERSE EVENTS:
Time Frame: 16 Weeks
Description: At entry, weeks 4,10, and 16, All-Cause Mortality and Serious Adverse Events were assessed.
Groups:
- 45 mg Daily: Participants in this arm take a daily 45 mg dose of zinc gluconate.
  Participants were interviewed for side effects at baseline and at week 16.
- 90 mg Daily: Participants in this arm take a daily 90 mg dose of zinc gluconate.
  Participants were interviewed for side effects at baseline and at week 16.
Arm/Group | 45 mg Daily | 90 mg Daily
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/27
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/27
Other Adverse Events (participants affected / at risk) | 0/25 | 1/27
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 45 mg Daily (N=25) | 90 mg Daily (N=27)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal cramps (Gastrointestinal disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Due to the small sample size and short study period, we cannot establish causation. We did not include a placebo control group for comparison. Our study focused on participants with treated HIV and documented zinc deficiency in the United States. We did not obtain dietary or physical activity patterns. Participants with treated HIV and documented zinc deficiency resided in the United States, therefore our findings cannot be generalized to different populations or to resource limited settings.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2016-12-08): https://cdn.clinicaltrials.gov/large-docs/69/NCT02856269/Prot_SAP_000.pdf
  • Informed Consent Form (2017-11-14): https://cdn.clinicaltrials.gov/large-docs/69/NCT02856269/ICF_001.pdf